CLINICAL TRIAL: NCT05911893
Title: the Effect of High Caloric Oral Nutritional Supplements on Growth and Development of Malnourished Children
Acronym: EHCONSGDMC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Collaborators: Anhui Provincial Children's Hospital (Other); Baoji Maternity and Child Healthcare Hospital (Unknown); Chengdu Women's and Children's Central Hospital (Other); Guiyang Maternity and Child Health Care Hospital (Other); Guangzhou Women and Children's Medical Center (Other); Hunan Children's Hospital (Other Government); Jiangxi Maternal and Child Health Hospital (Other); Kunming Children's Hospital (Other); Nanjing Maternity and Child Health Care Hospital (Other); Children's Hospital of The Capital Institute of Pediatrics (Other); Xianyang Children's Hospital (Other); Nestle Health Science (Industry); The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Chen Li, Associate Professor, Director, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHCONSGDMC
Record Dates: First submitted 2023-05-16; First posted 2023-06-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Malnutrition, Child; Malnourishment; Nutritional Deficiency; Undernutrition
Keywords: Oral Nutritional Supplements; Physique Growth; Neuropsychological Development
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition

STUDY DESIGN:
Intervention Model Description: Participants aged 1 to 3 years who are malnourished (underweight and wasting) are randomly divided into an experimental group and a control group. The experimental group is given nutritional education and high-energy total nutrition formula, while the control group is given nutritional education and dietary guidance. At the 1-month, 2-month, 3-month, and 6-month follow-ups of enrollment, children in the control group are transferred to the trial group if the assessment revealed that they are unable to achieve ≥75% of their predicted nutritional requirements through dietary modification or their rate of weight gain do not improve, according to the study design principles of the stepped wedge cluster trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high caloric oral nutritional supplements group (Experimental): Participants aged 1 to 3 years who are malnourished (underweight and wasting). They will receive nutritional education,dietary instruction and daily high caloric oral nutritional supplements for 12 months.
  Interventions: Dietary Supplement: high caloric oral nutritional supplements; Behavioral: nutritional education; Behavioral: dietary guidance
- nutritional education and dietary guidance group (Active Comparator): Participants aged 1 to 3 years who are malnourished (underweight and wasting). They will receive nutrition education and dietary instruction.
  Interventions: Behavioral: nutritional education; Behavioral: dietary guidance

INTERVENTIONS:
Dietary Supplement: high caloric oral nutritional supplements — High caloric oral nutritional supplements (which can supplement 30% of the energy requirement) is given daily, and the recommended amount of energy and protein is referred to the 2013 Chinese Dietary Nutrient Reference Intake Table. At 6 months of enrollment, participants will be asked to evaluate whether to continue feeding according to the experimental group protocol or to stop to ensure proper nutritional intake.
  Other Names: high-energy total nutrition formula
  Arms: high caloric oral nutritional supplements group
Behavioral: nutritional education — After enrollment,health education information is pushed approximately every 4 weeks through the WeChat platform or/and short text messages to parents.
Behavioral: dietary guidance — At follow-up visits at 0, 1, 2, 3, 6,and 12 months after enrollment, a professionally trained pediatrician give the participant's guardian dietary instructions appropriate to the age stage and physical condition of the child. Each session lasts approximately 10 minutes.

SUMMARY:
The goal of this clinical trial is to investigate the effect of high caloric oral nutritional supplements on body proportion, weight, linear growth pattern, neuropsychological development level and related health aspects (gut health, immune function, quality of life, etc.) in participants aged 1 to 3 years who are malnourished (underweight and wasting),as well as to evaluate the safety of applying high caloric oral nutritional supplements. Participants will receive nutritional education and daily high caloric oral nutritional supplements(experimental group),or will receive nutritional education and dietary instruction(control group).This study may provide data to support the development of clinical intervention strategies for malnourished Chinese children.

DETAILED DESCRIPTION:
Background:Growth and development is an important indicator of children's health and nutritional status, and nutrition is the most important material basis for growth and development. The prevention and treatment of malnutrition in children can be achieved by choosing whole nutritional formulas for special medical purposes as oral nutritional supplements (ONS), which has been confirmed by some overseas clinical studies to promote the growth benefit of malnourished children, but no multicenter clinical study has been conducted in China on the effect of ONS on the improvement of growth and development of malnourished Chinese children.

Objective and significance: To investigate the effects of high caloric ONS on body proportion, weight, linear growth pattern, neuropsychological development level and related health aspects (gut health, immune function, quality of life, etc.) in children, as well as to evaluate the safety of applying high caloric ONS, and to provide data to support the development of clinical intervention strategies for malnourished Chinese children.

Research design:A multicenter, randomized, controlled clinical trial design method is used to randomize children who meet the inclusion criteria into the experimental and control groups using a competitive entry method. The test group is given nutritional education and high caloric ONS (which can supplement 30% of the energy requirement), while the control group is given nutritional education and dietary instruction.Participants are followed up at 0, 1,2, 3, 6, and 12 months of enrollment. The investigators will collect dietary diaries, physical indicators, developmental quotient scores, quality of life measures, gut health, infectious disease-related questionnaires and safety indicators (blood biochemical indicators, urine routine) from children in both groups to comprehensively assess the effect of high caloric ONS intervention on physical growth, neuropsychological development levels and related aspects (gut health, immune function, quality of life, etc.) of malnourished children, as well as to conduct safety analyses.

Sample size:According to similar studies to date, a total of 200 people are recommended for this study.

Statistical analysis: Statistical analysis is performed using SAS 9.4. For continuous variables (height, weight, BMI-Z score, DQ score, etc.), statistical descriptions are performed using mean and standard deviation (conforming to normal distribution) or median and interquartile range (IQR); for categorical variables, statistical descriptions are performed using frequency and percentage; for the main efficacy indicators, mixed-effects models are used for efficacy evaluation indicators according to the principle of adjusted intentionality analysis (mITT). For the safety evaluation, the number, frequency and incidence of adverse events and reactions are calculated, and the positive abnormal changes of laboratory biochemical indexes such as blood routine, urine routine, liver and kidney function are counted. p value < 0.05 is considered statistically significant.

Ethical matters and data protection: The guardians of the children participating in the study will sign an informed consent form. This study is approved by the local ethics committee. Patients' names will be abbreviated and study data will be assigned a code which will then be provided to the investigator. Parental authorization for patient health information will remain in effect until the study is completed. After that, private information will be removed from the study records by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1-3 years
* BMI for Age Z-score<-2
* Height-for-age z score<-2
* Total daily energy intake<75% of recommended nutrient intake
* The child's guardian is willing to participate in this study and sign an informed consent form.

Exclusion Criteria:

* Chronic or severe infectious disease (e.g., chronic hepatitis, HIV or tuberculosis infection)
* Certain congenital or genetic diseases affecting physical growth and development (congenital heart disease, Down's syndrome, infantile anorexia nervosa, etc.), malignancies and use of drugs (diuretics, appetite stimulants, steroids and growth hormones, etc.)
* Severe gastrointestinal disorders (e.g., celiac disease, short bowel syndrome, inflammatory bowel disease, etc.)
* Acute and chronic respiratory/digestive tract infections within 2 weeks prior to enrollment
* Allergy or contraindication to any of the ingredients in the high-energy total nutrition formula used in this study
* Have used high-energy enteral nutrition preparations for the last 3 months

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
BMI for Age Z-score(BAZ) | at 6 months of enrollment
  Trained research assistants or health care practitioners obtain weight in kilograms and height in centimeters (mean of 3 consecutive measurements). Height and weight will be combined to report BMI in kg/m^2.Then, the BAZ is calculated using WHO2011v3.2.2 software.

SECONDARY OUTCOMES:
Dietary Diary | at 0, 1, 2, 3, 6 and 12 months of enrollment
  Participants provide a dietary diary over an average two-day period through a WeChat app each visit. The app prompts participants to record and estimate details of all meals and snacks they consumed, especially formula used in the study.
BMI for Age Z-score(BAZ) | at 0, 1, 2, 3 and 12 months of enrollment
  Trained research assistants or health care practitioners obtain weight in kilograms and height in centimeters (mean of 3 consecutive measurements). Height and weight will be combined to report BMI in kg/m^2.Then, the BAZ is calculated using WHO2011v3.2.2 software.
Weight for Age Z-score(WAZ) | at 0, 1, 2, 3, 6 and 12 months of enrollment
  Trained research assistants or health care practitioners obtain weight in kilograms using a standardized approach. Weight is measured using a precision digital scale or mechanical scale(mean of 3 consecutive measurements). Then, the WAZ is calculated using WHO2011v3.2.2 software.
Height for Age Z-score(HAZ) | at 0, 1, 2, 3, 6 and 12 months of enrollment
  Trained research assistants or health care practitioners obtain height in centimeters using a standardized approach. Height is measured with a calibrated stadiometer(mean of 3 consecutive measurements). Then, the HAZ is calculated using WHO2011v3.2.2 software.
Gesell Developmental Scale Test | at 0, 6, and 12 months of enrollment
  Mainly assesses participants in 5 areas:adaptive behavior, gross motor, fine motor, language behavior,personal-social behavior, the evaluation finally calculates the developmental quotient (DQ) of each area. Diagnostic criteria: DQ is more than or equal to 86 is normal, DQ is marginal between 76 and 85, DQ is mild mental retardation between 55 and 75, DQ is moderate mental retardation between 40 and 54, DQ is severe mental retardation between 25 and 39, and DQ is less than or equal to 25 is extremely severe mental retardation.
Infants - Junior High School Students Social Competence Test (S-M test) | at 0, 6, and 12 months of enrollment
  The scale, derived from the revised version of the Japanese Social Competence test (S-M test) and revised by a Chinese researcher, is applicable to children from 6 months of age to 14 years of age and includes 132 items in 6 sections with 7 starting ages, which are filled in item by item by parents or daily caregivers according to the appropriate age, with ≥10 being normal.
Pediatric Quality of Life Inventory (PedsQL) | at 0, 6, and 12 months of enrollment
  The quality of life of the participants is assessed using the Pediatric Quality of Life Inventory.The Infant Scale or Generic Core Scales is completed according to age.Scores are transformed on a scale from 0 to 100,with higher scores indicating better quality of life.
the Chinese version of the World Health Organization Quality of Life-BREF (WHOQOL-BREF) | at 0, 6 and 12 months of enrollment
  The quality of life of parents is assessed using the WHOQOL-BREF.The WHOQOL-BREF, comprises 26 items, two general items and 24 others, across the following four domains: physical (7 items), psychological (6 items), social (3 items), and environmental (8 items).Calculate the average score of all items in each domain, converted into a score of 4 to 20 or 0 to100 by two algorithms,with higher scores indicating better quality of life.
Gut Health Questionnaire | at 0, 1，3, 6, and 12 months of enrollment
  A questionnaire is used to understand gut health, including entries on the Bristol Stool Scale (to assess stool status), the average number of bowel movements per day, and the frequency of bloating and abdominal pain.
Infectious Diseases Related Questionnaire | at 0, 1，3, 6, and 12 months of enrollment
  A infectious disease-related questionnaire is used to understand immune function, including the number and duration of upper respiratory tract infections, infectious diarrhea.
Blood Routine Test | at 0, 6 and 12 months of enrollment
  Blood routine test is completed at 0, 6 and 12 months of enrollment for safety analysis.Includes the following parameters:white blood cell count,red blood cell count,hemoglobin,mean corpuscular hemoglobin concentration,platelet,standard deviation in red cell distribution width,coefficient variation of red blood cell volume distribution width,platelet distribution width,mean platelet volume,platelet larger cell ratio,thrombocytocrit,neutrophil ratio,lymphocyte ratio,monocyte ratio,eosinophil ratio,basophil ratio,neutrophil count,lymphocyte count,monocyte count,eosinophil count,basophil count.
Liver Function Test | at 0, 6 and 12 months of enrollment
  Liver function test is completed at 0, 6 and 12 months of enrollment for safety analysis.Includes the following parameters:total protein,albumin,globulin,alanineamino transferase,aspartate amino transferase,bilirubin,direct bilirubin,total bile acid,alkaline phosphatase,amma-glutamyl transpeptidase.
Renal Function Test | at 0, 6 and 12 months of enrollment
  Renal function test is completed at 0, 6 and 12 months of enrollment for safety analysis.Includes the following parameters:creatinine,blood urea nitrogen.
Urine Routine Test | at 0, 6 and 12 months of enrollment
  Urine routine test is completed at 0, 6 and 12 months of enrollment for safety analysis.Includes the following parameters:urinary bilirubin,urinary ketone bodies,blood,urinary white blood cells,urinary red blood cells,urinary sugar,urinary protein,urinary cast.

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen, doctor, Study Director — Children's Hospital of Chongqing Medical University
Locations (13):
- China (13):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - Children's Hospital of The Capital Institute of Pediatrics, Beijing, Beijing Municipality
  - The First Hospital of Jilin University, Jilin, Changchun
  - Growth, Development and Mental health of Children and Adolescence Center, Chongqing, Chongqing Municipality
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Guiyang Maternity and Child Health Care Hospital, Guiyang, Guizhou
  - Hunan Children's Hospital, Changsha, Hunan
  - Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Baoji Maternity and Child Healthcare Hospital, Baoji, Shanxi
  - Xianyang Children's Hospital, Xianyang, Shanxi
  - Chengdu Women's and Children's Central Hospital，School of Medicine，University of Electronic Science and Technology of China, Chengdu, Sichuan
  - Kunming Children's Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No
Data is confidential during the study.

REFERENCES:
- [Background] Hemming K, Taljaard M, McKenzie JE, Hooper R, Copas A, Thompson JA, Dixon-Woods M, Aldcroft A, Doussau A, Grayling M, Kristunas C, Goldstein CE, Campbell MK, Girling A, Eldridge S, Campbell MJ, Lilford RJ, Weijer C, Forbes AB, Grimshaw JM. Reporting of stepped wedge cluster randomised trials: extension of the CONSORT 2010 statement with explanation and elaboration. BMJ. 2018 Nov 9;363:k1614. doi: 10.1136/bmj.k1614. PMID 30413417